CLINICAL TRIAL: NCT00123201
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Efficacy, Safety and Tolerability Study of Dronabinol MDI in the Acute Treatment of Migraine Headache
Brief Title: Study to Evaluate the Efficacy and Safety of Dronabinol Metered Dose Inhaler (MDI) in Acute Treatment of Migraine Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: Nektar Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S175.2.103
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2006-09

CONDITIONS: Migraine With Aura; Migraine Without Aura
Keywords: efficacy & safety, migraine headache, placebo-controlled; migraine headache with or without aura
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Migraine Disorders

INTERVENTIONS:
Drug: Dronabinol MDI

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of dronabinol MDI for the acute treatment of moderate to severe migraine headache.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 to 65 years, inclusive, with clinically diagnosed migraine with or without aura based on International Headache Society criteria

Exclusion Criteria:

* Subjects who experience migraine with prolonged aura; familiar hemiplegic migraine; migrainous infarction or basilar migraine; and those with greater than eight migraine attacks per month and/or greater than 14 migraine days per month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (29):
- United States (29):
  - Site 10, Huntsville, Alabama
  - Site 8, Huntsville, Alabama
  - Site 11, Tucson, Arizona
  - Site 3, Anaheim, California
  - Site 6, San Francisco, California
  - Site 15, Stockton, California
  - Site 26, Melbourne, Florida
  - Site 22, New Port Richey, Florida
  - Site 18, Orange City, Florida
  - Site 27, Pembroke Pines, Florida
  - Site 14, Plantation, Florida
  - Site 24, Plantation, Florida
  - Site 7, St. Petersburg, Florida
  - Site 25, Atlanta, Georgia
  - Site 12, Chicago, Illinois
  - Site 1, Chicago, Illinois
  - Site 28, Lexington, Kentucky
  - Site 20, Madisonville, Kentucky
  - Site 2, Boston, Massachusetts
  - Site 19, Omaha, Nebraska
  - Site 29, Clementon, New Jersey
  - Site 4, Mount Vernon, New York
  - Site 9, Raleigh, North Carolina
  - Site 23, Fargo, North Dakota
  - Site 13, Portland, Oregon
  - Site 5, Spartanburg, South Carolina
  - Site 16, Bryan, Texas
  - Site 17, Colleyville, Texas
  - Site 21, Alexandria, Virginia